CLINICAL TRIAL: NCT04411082
Title: A Phase 2 Study to Evaluate the Safety and Tolerability of IMR-687 in Subjects With Beta Thalassemia
Brief Title: A Study of IMR-687 in Subjects With Beta Thalassemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IMR-BTL-201demonstrated that while IMR-687 was generally well-tolerated, it failed to show any meaningful benefit in transfusion burden or improvement in most disease-related biomarkers. So, the sponsor has decided to discontinue this study
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Collaborators: Imara, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMR-BTL-201; 2019-002989-12 (EudraCT Number)
Record Dates: First submitted 2020-04-15; First posted 2020-06-02 (Actual); Results first posted 2022-06-30 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: β Thalassemia
Keywords: Transfusion; TDT; NTDT

STUDY DESIGN:
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lower Dose IMR-687 (Experimental): Oral administration of once daily IMR-687
  Interventions: Drug: IMR-687
- Higher dose IMR-687 (Experimental): Oral administration of once daily IMR-687
  Interventions: Drug: IMR-687
- Placebo (Placebo Comparator): Oral administration of once daily placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMR-687 — Oral administration of once daily IMR-687
  Arms: Higher dose IMR-687; Lower Dose IMR-687
Drug: Placebo — Oral administration of once daily Placebo
  Arms: Placebo

SUMMARY:
A Study to Evaluate the Safety and Tolerability of IMR-687 in Subjects with Beta Thalassemia

DETAILED DESCRIPTION:
A phase 2, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK, and PD of IMR-687 (phosphodiesterase (PDE) 9 inhibitor) administered once daily (qd) orally for 36 weeks in 2 populations of adult subjects with β-thalassemia: Population 1 (Transfusion Dependent Thalassemia (TDT) subjects) and Population 2 (Non-Transfusion Dependent Thalassemia (NTDT) subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of β-thalassemia or HbE/ β-thalassemia in their medical history. Concomitant alpha gene deletion, duplication, or triplication is allowed.
2. Documentation of the dates of transfusion events and the number of all pRBC units per event within the 12 weeks prior to the Baseline (Day 1) visit. .
3. Must be willing and able to complete all study assessments and procedures, and to communicate effectively with the investigator and site staff.
4. TDT Subjects: subjects must be regularly transfused, defined as >3 to 10 pRBC units in the12 weeks prior to Baseline (Day 1) visit and no transfusion-free period for >35 days during that period.
5. NTDT subjects: Subjects must be transfusion independent, defined as 0 to ≤3 units of pRBCs received during the 12-week period prior to the Baseline (Day 1) visit, must not be on a regular transfusion program, must be RBC transfusion-free for at least ≥ 4 weeks prior to randomization, and must not be scheduled to start a regular
6. hematopoietic stem cell transplantation within 9 months.
7. NTDT subjects: Subjects must have Hb ≤10.0 g/dL at Screening; the screening Hb sample must be collected 7 to 28 days prior to randomization. Hb values within 21 days post-transfusion will be excluded.
8. ECOG performance score of 0 to 1
9. Female subjects must not be pregnant, or breastfeeding and be highly unlikely to become pregnant. Male subjects must be unlikely to impregnate a partner.

Exclusion Criteria:

1. Diagnosis of α-thalassemia (e.g., hemoglobin H [HbH]) or hemoglobin S (HbS)/ β thalassemia.
2. Body mass index (BMI) <17.0 kg/m2 or a total body weight <45 kg; or BMI >35 kg/m2
3. Subjects with known active hepatitis A, hepatitis B, or hepatitis C, with active or acute event of malaria, or who are known to be positive for human immunodeficiency virus (HIV).
4. Stroke requiring medical intervention ≤24 weeks prior to randomization.
5. Platelet count >1000 × 109/L.
6. Participated in another clinical study of an investigational agent (or device) within 30 days or 5-half-lives of date of informed consent, whichever is longer, or is currently participating in another study.
7. For Subjects on iron chelation therapy (ICT) at the time of ICF signing, initiation of ICT less than 24 weeks before the predicted randomization date.
8. Prior exposure to sotatercept or luspatercept, IMR-687, or gene therapy within 6 months prior to randomization (Day 1).
9. Subjects who have major organ damage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Luperchio, Study Director — Cardurion Pharmaceuticals
Locations (36):
- Herlev Hospital, Herlev, Capital Region, Denmark
- France (3):
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse, Haute-Garonn
  - Hôpital Edouard Herriot, Lyon, Rhone
  - Hôpital Necker-Enfants Malades, Paris
- Georgia (3):
  - M. Zodelava Hematology Centre, Tbilisi, Borjomi
  - National Center of Surgery, Tbilisi
  - Medinvest - Institute of Hematology and Transfusiology, Tbilisi
- Greece (4):
  - Aghia Sofia General Children's Hospital, Athens, Attica
  - Laiko General Hospital of Athens, Athens, Attica
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki, Central Macedonia
  - University General Hospital of Patras, Patra, Peloponnese
- Israel (4):
  - Rambam Health Care Campus, Haifa, Haifa District
  - Hadassah University Hospital Ein Kerem, Jerusalem, Jerusalem
  - The Galilee Medical Center, Nahariya, Northern District
  - Emek Medical Center, Afula
- Italy (2):
  - Azienda Ospedaliera Giuseppe Brotzu, Orbassano, Turin
  - Azienda Ospedaliera Universitaria - Università degli Studi della Campania Luigi Vanvitelli, Orbassano, Turin
- Chronic Care Center, Hazmiyeh, Lebanon
- Malaysia (6):
  - Hospital Sultanah Aminah Johor Bharu, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Queen Elizabeth - Kota Kinabalu, Kota Kinabalu, Sabah
  - Hospital Umum Sarawak, Kuching, Sarawak
- Hôpital d'Enfants Rabat, Rabat, Morocco
- Amsterdam Universitair Medische Centra - Academisch Medisch Centrum, Amsterdam, North Holland, Netherlands
- Tunisia (3):
  - Centre Hôpital Universitaire Farhat Hached, Sousse
  - Centre National de Greffe de la Moelle Osseuse, Tunis
  - Hospital Aziza Othmana, Tunis
- Turkey (Türkiye) (4):
  - Akdeniz Üniversitesi, Mersin, Mersin
  - Mersin Üniversitesi Tıp Fakültesi, Mersin, Mersin
  - Hacettepe Üniversitesi, Ankara
  - Ege Universitesi Tip Fakultesi, Izmir
- United Kingdom (3):
  - Whittington Health NHS Trust, London, England
  - University College London Hospitals NHS Foundation Trust, London, England
  - Manchester University NHS Foundation Trust, Manchester, England

REFERENCES:
- [Derived] Foong WC, Loh CK, Ho JJ, Lau DS. Foetal haemoglobin inducers for reducing blood transfusion in non-transfusion-dependent beta-thalassaemias. Cochrane Database Syst Rev. 2023 Jan 13;1(1):CD013767. doi: 10.1002/14651858.CD013767.pub2. PMID 36637054

RESULTS

PARTICIPANT FLOW:
Groups:
- TDT High Dose: TDT High dose
- TDT Low Dose: TDT Low dose
- TDT Placebo: TDT Placebo
- NTDT High Dose: NTDT High dose
- NTDT Low Dose: NTDT Low dose
- NTDT Placebo: NTDT Placebo
Period: Overall Study
Arm/Group | TDT High Dose | TDT Low Dose | TDT Placebo | NTDT High Dose | NTDT Low Dose | NTDT Placebo
Started | 29 | 25 | 20 | 24 | 12 | 12
Completed | 18 | 16 | 16 | 10 | 8 | 6
Not Completed | 11 | 9 | 4 | 14 | 4 | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | TDT High Dose | TDT Low Dose | TDT Placebo | NTDT High Dose | NTDT Low Dose | NTDT Placebo | Total
Number analyzed (Participants) | 29 | 25 | 20 | 24 | 12 | 12 | 122
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (12.06) | 30.0 (9.95) | 31.3 (8.57) | 34.1 (12.64) | 28.5 (8.21) | 36.0 (9.56) | 31.9 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 9 | 10 | 6 | 8 | 63
  Male | 14 | 10 | 11 | 14 | 6 | 4 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 7 | 4 | 4 | 3 | 4 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1 | 0 | 2
  White | 19 | 17 | 14 | 17 | 7 | 6 | 80
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 2 | 3 | 1 | 2 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 1 | 0 | 0 | 2 | 0 | 1 | 4
  Malaysia | 4 | 6 | 4 | 3 | 3 | 2 | 22
  Greece | 9 | 2 | 1 | 5 | 0 | 2 | 19
  Lebanon | 0 | 4 | 3 | 0 | 1 | 0 | 8
  Netherlands | 0 | 0 | 0 | 2 | 0 | 1 | 3
  Turkey | 3 | 5 | 7 | 1 | 0 | 0 | 16
  Morocco | 1 | 1 | 0 | 2 | 0 | 2 | 6
  Denmark | 3 | 0 | 2 | 0 | 0 | 0 | 5
  Italy | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Georgia | 0 | 2 | 1 | 3 | 1 | 1 | 8
  Israel | 2 | 2 | 2 | 1 | 0 | 0 | 7
  France | 2 | 1 | 0 | 0 | 2 | 2 | 7
  Tunisia | 4 | 2 | 0 | 5 | 4 | 0 | 15
BMI [Mean (Standard Deviation); unit: kg/m2] | 22.900 (3.2252) | 21.252 (2.2874) | 22.699 (2.9968) | 22.031 (3.5415) | 21.1320 (3.5047) | 21.9120 (3.5638) | 22.0873 (3.1573)
Serum Ferritin [Mean (Standard Deviation); unit: micrograms per liter] | 1724.4 (1857.66) | 3449.1 (5093.24) | 1793.3 (1844.72) | 981.4 (951.29) | 945.8 (962.09) | 447.8 (222.32) | 1726.69 (2740.18)

OUTCOME MEASURES:

1. Primary Outcome: IMR-687 Safety and Tolerability
Description: Incidence and severity of Adverse Events Incidence and severity of Serious Adverse Events
Time Frame: Baseline to Week 40
Population: Safety Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | TDT High Dose | TDT Low Dose | TDT Placebo | NTDT High Dose | NTDT Low Dose | NTDT Placebo
Number analyzed (Participants) | 29 | 25 | 20 | 24 | 12 | 12
Participants
  Treatment emergent Adverse Events | 25 | 22 | 15 | 18 | 12 | 6
  Treatment emergent Adverse Event related to study drug | 19 | 15 | 8 | 11 | 7 | 4
  Grade 3 or greater treatment emergent Adverse Event | 4 | 9 | 2 | 4 | 1 | 1

2. Secondary Outcome: TDT Patients: Reduction in Red Blood Cell (RBC) Transfusion Burden With ≥33% Hematological Improvement From Week 12 to Week 24
Description: Proportion of patients with ≥33% hematological improvement (as measured by reduced transfusion burden) from Week 12 to Week 24 compared to the 12 weeks prior to Baseline (Day 1)
Time Frame: Baseline to Week 24
Population: Per Protocol Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TDT High Dose | TDT Low Dose | TDT Placebo
Number analyzed (Participants) | 21 | 18 | 18
Participants | 2 | 1 | 2
Statistical Analysis 1: Comparison: TDT High Dose vs TDT Low Dose vs TDT Placebo; Test type: Superiority; p > 0.99, Fisher Exact

3. Secondary Outcome: NTDT Patients: Proportion of Subjects With an Increase From Baseline of Hb at Week 12 to Week 24 in the Absence of Transfusions.
Description: Proportion of subjects with an increase from baseline of ≥1.0 g/dL in mean Hb values at Week 12 to Week 24 in the absence of transfusions.
Time Frame: Baseline to Week 24
Population: Per protocol analysis
Measure: Count of Participants; unit: Participants
Arm/Group | NTDT High Dose | NTDT Low Dose | NTDT Placebo
Number analyzed (Participants) | 15 | 10 | 10
Participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: NTDT High Dose vs NTDT Low Dose vs NTDT Placebo; Test type: Superiority; p > 0.99, Fisher Exact

4. Secondary Outcome: NTDT Patients: Proportion of Subjects With an Increase From Baseline of ≥3% in Mean HbF Values at Week 12 to Week 24 in Absence of Transfusions
Description: Proportion of subjects with an increase from baseline of ≥3% in mean HbF values at Week 12 to Week 24 in absence of transfusions
Time Frame: Baseline to Week 24
Population: Per Protocol Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | NTDT High Dose | NTDT Low Dose | NTDT Placebo
Number analyzed (Participants) | 11 | 5 | 8
Participants | 1 | 1 | 0
Statistical Analysis 1: Comparison: NTDT High Dose vs NTDT Low Dose vs NTDT Placebo; Test type: Superiority; p > 0.99, Fisher Exact

5. Secondary Outcome: TDT Patients: Reduction in Red Blood Cell (RBC) Transfusion Burden With ≥33% Hematological Improvement From Week 24 to Week 36
Description: Proportion of patients with ≥33% hematological improvement from Week 24 to Week 36 compared to the 12 weeks prior to Baseline (Day 1)
Time Frame: Baseline to Week 36
Population: Per Protocol Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TDT High Dose | TDT Low Dose | TDT Placebo
Number analyzed (Participants) | 16 | 13 | 15
Participants | 0 | 1 | 1
Statistical Analysis 1: Comparison: TDT High Dose vs TDT Low Dose vs TDT Placebo; Test type: Superiority; p > 0.4839, Fisher Exact

6. Secondary Outcome: TDT Patients: Reduction in Red Blood Cell (RBC) Transfusion Burden With ≥50 % Hematological Improvement From Week 12 to Week 24
Description: Proportion of patients with ≥50% hematological improvement from Week 12 to Week 24 compared to the 12 weeks prior to Baseline (Day 1)
Time Frame: Baseline to Week 24
Population: Per Protocol Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TDT High Dose | TDT Low Dose | TDT Placebo
Number analyzed (Participants) | 21 | 18 | 18
Participants | 0 | 0 | 2
Statistical Analysis 1: Comparison: TDT High Dose vs TDT Low Dose vs TDT Placebo; Test type: Superiority; p = 0.2065, Fisher Exact

7. Secondary Outcome: TDT Patients: Reduction in Red Blood Cell (RBC) Transfusion Burden With ≥50% Hematological Improvement From Week 24 to Week 36
Description: Proportion of patients with ≥50% hematological improvement from Week 24 to Week 36 compared to the 12 weeks prior to Baseline (Day 1)
Time Frame: Baseline to Week 36
Population: Per Protocol Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TDT High Dose | TDT Low Dose | TDT Placebo
Number analyzed (Participants) | 16 | 13 | 15
Participants | 0 | 1 | 1
Statistical Analysis 1: Comparison: TDT High Dose vs TDT Low Dose vs TDT Placebo; Test type: Superiority; p = 0.4839, Fisher Exact

8. Secondary Outcome: NTDT Patients: Proportion of Subjects With an Increase From Baseline of Hb at Week 24 to Week 36 in the Absence of Transfusions
Description: Proportion of subjects with an increase from baseline of ≥1.0 g/dL in mean Hb values at Week 24 to Week 36 in the absence of transfusions.
Time Frame: Baseline to Week 36
Population: Per Protocol Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | NTDT High Dose | NTDT Low Dose | NTDT Placebo
Number analyzed (Participants) | 12 | 9 | 8
Participants | 1 | 1 | 0
Statistical Analysis 1: Comparison: NTDT High Dose vs NTDT Low Dose vs NTDT Placebo; Test type: Superiority; p > 0.99, Fisher Exact

9. Secondary Outcome: NTDT: Proportion of Subjects With an Increase From Baseline of ≥3% in Mean HbF Values at Week 24 to Week 36 in Absence of Transfusions
Description: Proportion of subjects with an increase from baseline of ≥3% in mean HbF values at Week 24 to Week 36 in absence of transfusions
Time Frame: Baseline to Week 36
Population: Per Protocol Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | NTDT High Dose | NTDT Low Dose | NTDT Placebo
Number analyzed (Participants) | 8 | 6 | 7
Participants | 1 | 0 | 0
Statistical Analysis 1: Comparison: NTDT High Dose vs NTDT Low Dose vs NTDT Placebo; Test type: Superiority; p > 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | TDT High Dose | TDT Low Dose | TDT Placebo | NTDT High Dose | NTDT Low Dose | NTDT Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/25 | 0/20 | 0/24 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/29 | 3/25 | 1/20 | 3/24 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 25/29 | 22/25 | 15/20 | 18/24 | 12/12 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDT High Dose (N=29) | TDT Low Dose (N=25) | TDT Placebo (N=20) | NTDT High Dose (N=24) | NTDT Low Dose (N=12) | NTDT Placebo (N=12)
Carbon Monoxide Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDT High Dose (N=29) | TDT Low Dose (N=25) | TDT Placebo (N=20) | NTDT High Dose (N=24) | NTDT Low Dose (N=12) | NTDT Placebo (N=12)
Headache (Nervous system disorders) | 10 | 10 | 7 | 5 | 2 | 2
Nausea (Gastrointestinal disorders) | 11 | 6 | 1 | 5 | 1 | 1
Dizziness (Nervous system disorders) | 5 | 5 | 2 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 2 | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 3 | 2 | 0
Vomitting (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 2 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 2 | 1
COVID19 (Infections and infestations) | 1 | 3 | 0 | 3 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT04411082/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT04411082/SAP_001.pdf